CLINICAL TRIAL: NCT01654211
Title: A Three-Part Study Evaluating the Pharmacokinetics of Intravenous (IV) Danoprevir (DNV)/Oral Low-Dose Ritonavir (RTV), the Absolute Bioavailability of DNV With and Without Oral Low-Dose RTV, and the Effect of Oral Cyclosporine on IV DNV/Oral Low-Dose RTV in Healthy Adult Volunteers
Brief Title: A Pharmacokinetic And Bioavailability Study of Intravenous Danoprevir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: NP28297; 2012-000470-40 (EudraCT Number)
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Ritonavir

STUDY DESIGN:
Who Masked: Participant

ARMS (7):
- Part 1: iv danoprevir (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir
- Part 1: placebo (Placebo Comparator)
  Interventions: Drug: placebo; Drug: ritonavir
- Part 2 A: iv danoprevir (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir
- Part 2 B: oral danoprevir (Active Comparator)
  Interventions: Drug: danoprevir; Drug: ritonavir
- Part 2 C: ritonavir (Active Comparator)
  Interventions: Drug: ritonavir
- Part 3 D: iv danoprevir (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir
- Part 3 E: iv danoprevir + cyclosporine (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — single iv infusion
  Arms: Part 1: iv danoprevir; Part 2 A: iv danoprevir; Part 3 D: iv danoprevir; Part 3 E: iv danoprevir + cyclosporine
Drug: danoprevir — single oral dose
  Arms: Part 2 B: oral danoprevir
Drug: placebo — single iv infusion
  Arms: Part 1: placebo
Drug: ritonavir — oral doses

SUMMARY:
This three-part study will evaluate the pharmacokinetics and bioavailability of intravenous danoprevir with and without low-dose oral ritonavir, and the effect of oral cyclosporine on the pharmacokinetics of intravenous danoprevir with ritonavir in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy male and female nonsmoking volunteers, 18 to 55 years of age inclusive; healthy status will be defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history and a complete physical examination

Exclusion Criteria:

* Pregnant or lactating women or males with female partners who are pregnant or lactating
* Positive results for drugs of abuse at screening or prior to admission to the clinical site during any study period
* Positive for hepatitis B, hepatitis C or HIV infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve (AUC) | Pre-dose and up to 12 hours post-dose
Safety: Incidence of adverse events | approximately 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands